CLINICAL TRIAL: NCT02030782
Title: Youth Partners in Care: Depression & Quality Improvement
Brief Title: Youth Partners in Care: Depression and Quality Improvement
Acronym: YPIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Collaborators: RAND (Other); Kaiser Permanente (Other); University of Pittsburgh (Other); Venice Family Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HS009908
Record Dates: First submitted 2012-01-19; First posted 2014-01-09 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2008-12

CONDITIONS: Depression
Keywords: depression; quality improvement; treatment; adolescents
MeSH Terms: conditions — Depression | interventions — Quality Improvement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (Active Comparator): Patients received usual care through primary care, enhanced by provider education regarding depression evaluation and management (1-2 hour training, plus study manual)
  Interventions: Other: Usual Care
- Quality Improvement for Depression (Experimental): Major intervention components included a) expert leader teams who planned and implemented the intervention at each clinic, b) care managers who supported primary care clinicians with depression evaluation and management, c) access to cognitive-behavior therapy for depression within each primary care clinic, and d) patient and provider choice regarding treatment modality.
  Interventions: Other: Quality Improvement (QI) for depression

INTERVENTIONS:
Other: Quality Improvement (QI) for depression — Major intervention components included a) expert leader teams who planned and implemented the intervention at each clinic, b) care managers who supported primary care clinicians with depression evaluation and management, c) access to cognitive-behavior therapy for depression within each primary care clinic, and d) patient and provider choice regarding treatment modality.
  Arms: Quality Improvement for Depression
Other: Usual Care — Usual care enhanced by provider education regarding depression evaluation and management
  Arms: Usual Care

SUMMARY:
This randomized effectiveness trial evaluates a quality improvement intervention aimed at providing access to evidence-based depression treatments (particularly cognitive-behavior therapy for depression and or pharmacotherapy) through primary care for youth ages 13-21, as compared to enhanced usual care. The major hypothesis is that the quality improvement intervention will be associated with improved outcomes, relative to enhanced usual care.

ELIGIBILITY:
Inclusion Criteria:

* Met either of two criteria: 1) endorsed "stem items" for major depression or dysthymia from the 12-month Composite International Diagnostic Interview(CIDI-12,2.1) modified slightly to conform to diagnostic criteria for adolescents, 1-week or more of past-month depressive symptoms, and a total Center for Epidemiological Studies- Depression Scale(CES-D)40 score ≥ 16, or 2) CES-D score ≥ 24.
* Age 13-21
* Presented at primary care clinic

Exclusion Criteria:

* not English-speaking
* provider not in study
* sibling already in study
* completed eligibility screener previously

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 418 (Actual)
Dates: Start 1999-10; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Self-reported depressive symptoms on the CES-D (Center for Epidemiologic Studies Depression Scale) | 6-months

SECONDARY OUTCOMES:
mental health related quality of life as assessed using self-report on the Medical Outcomes Study Short Form 12 Health Survey. | 6 months, with follow up at 12 and 18 months
satisfaction with care | 6 months with follow up at 12 and 18 months
Rates of mental health care, counseling/psychotherapy, and medication treatment. | 6-months with follow-up at 12 and 18 months
  Youth self report on the study version of the Service Assessment for Children & Adolescents provided measures of rates of mental health care(dichotomous indicator of whether any mental health treatment received), counseling/psychotherapy (dichotomous indicator of whether counseling/psychotherapy was received, number of counseling/psychotherapy sessions), and medication treatment (dichotomous indicator of whether youth received any medication treatment for mental health problems). These measures were obtained using .

CONTACTS AND LOCATIONS:
Overall Officials: Joan R Asarnow, PhD, Principal Investigator — University of California, Los Angeles
Locations (5):
- United States (5):
  - University of California, Los Angeles, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Venice Family Clinic, Venice, California
  - Ventura County Medical Center, Ventura, California
  - University of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Asarnow JR, Jaycox LH, Anderson M. Depression among youth in primary care models for delivering mental health services. Child Adolesc Psychiatr Clin N Am. 2002 Jul;11(3):477-97, viii. doi: 10.1016/s1056-4993(02)00006-8. PMID 12222079
- [Background] Wells KB, Kataoka SH, Asarnow JR. Affective disorders in children and adolescents: addressing unmet need in primary care settings. Biol Psychiatry. 2001 Jun 15;49(12):1111-20. doi: 10.1016/s0006-3223(01)01113-1. PMID 11430853
- [Result] Asarnow JR, Jaycox LH, Tang L, Duan N, LaBorde AP, Zeledon LR, Anderson M, Murray PJ, Landon C, Rea MM, Wells KB. Long-term benefits of short-term quality improvement interventions for depressed youths in primary care. Am J Psychiatry. 2009 Sep;166(9):1002-10. doi: 10.1176/appi.ajp.2009.08121909. Epub 2009 Aug 3. PMID 19651711
- [Result] Asarnow JR, Jaycox LH, Duan N, LaBorde AP, Rea MM, Murray P, Anderson M, Landon C, Tang L, Wells KB. Effectiveness of a quality improvement intervention for adolescent depression in primary care clinics: a randomized controlled trial. JAMA. 2005 Jan 19;293(3):311-9. doi: 10.1001/jama.293.3.311. PMID 15657324
- [Result] Jaycox LH, Asarnow JR, Sherbourne CD, Rea MM, LaBorde AP, Wells KB. Adolescent primary care patients' preferences for depression treatment. Adm Policy Ment Health. 2006 Mar;33(2):198-207. doi: 10.1007/s10488-006-0033-7. PMID 16502131
- [Result] Asarnow JR, Jaycox LH, Duan N, LaBorde AP, Rea MM, Tang L, Anderson M, Murray P, Landon C, Tang B, Huizar DP, Wells KB. Depression and role impairment among adolescents in primary care clinics. J Adolesc Health. 2005 Dec;37(6):477-83. doi: 10.1016/j.jadohealth.2004.11.123. PMID 16310125
- [Result] Ngo VK, Asarnow JR, Lange J, Jaycox LH, Rea MM, Landon C, Tang L, Miranda J. Outcomes for youths from racial-ethnic minority groups in a quality improvement intervention for depression treatment. Psychiatr Serv. 2009 Oct;60(10):1357-64. doi: 10.1176/ps.2009.60.10.1357. PMID 19797376
- [Result] Tang L, Duan N, Klap R, Asarnow JR, Belin TR. Applying permutation tests with adjustment for covariates and attrition weights to randomized trials of health-services interventions. Stat Med. 2009 Jan 15;28(1):65-74. doi: 10.1002/sim.3453. PMID 18937226
- [Result] Goldstein RB, Asarnow JR, Jaycox LH, Shoptaw S, Murray PJ. Correlates of "non-problematic" and "problematic" substance use among depressed adolescents in primary care. J Addict Dis. 2007;26(3):39-52. doi: 10.1300/J069v26n03_05. PMID 18018807
- [Result] Fordwood SR, Asarnow JR, Huizar DP, Reise SP. Suicide attempts among depressed adolescents in primary care. J Clin Child Adolesc Psychol. 2007 Jul-Sep;36(3):392-404. doi: 10.1080/15374410701444355. PMID 17658983